CLINICAL TRIAL: NCT02561351
Title: Correlation Between Fractional Exhaled Nitric Oxide (FeNO) Levels and Asthma Exacerbation
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Mahidol University, Mahidol University
Other Study IDs: Si237/2013
Record Dates: First submitted 2015-09-16; First posted 2015-09-28 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Bronchial Asthma
Keywords: bronchial asthma; fractional exhaled nitric oxide (FeNO); asthma exacerbation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: FeNO measurement — FeNO was performed repeatedly every 3 months in every cases. exacerbations were recorded each visit

SUMMARY:
The purpose of this study is to determine mean or median of fractional exhaled nitric oxide (FeNO) in Thai atopic asthmatic children that divided into subgroups due to asthma exacerbation according to the global initiative for asthma guideline.

DETAILED DESCRIPTION:
From many previous studies, fractional exhaled nitric oxide (FeNO) has many benefits such as non-invasive, easily to perform, less time consume, has direct association with severity of inflammation of bronchial trees and sputum eosinophils, has benefit for diagnosis and monitoring the treatment in asthmatic patients.

In Thailand, this field of study is less extend, especially in children population. The investigators hypothesized that patients with asthma exacerbation may have high level of fractional exhaled nitric oxide (FeNO) than non exacerbation group.

It is therefore desirable to examine the association between fractional exhaled nitric oxide (FeNO) and asthma exacerbation among atopic asthmatic Thai children and will be the main objective of this research.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of atopic bronchial asthma follow up in clinic of allergy and clinical immunology, Siriraj hospital

Exclusion Criteria:

* smoker or past history of smoking
* chronic disease eg. HIV infection, pulmonary hypertension, systemic lupus erythematosus, liver cirrhosis, gastroesophageal reflux, COPD, bronchiectasis
* drink ethanol within 48 hours before enrollment
* history of upper or lower respiratory tract infection within 6 weeks before enrollment drink caffeine within day before enrollment during pregnancy history of systemic steroid use within 8 weeks before enrollment

Ages: 7 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: atopic asthmatic patients in Department of Pediatrics, Siriraj hospital (tertiary care)
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of asthma exacerbation in the studied cases with different FeNO levels | 1 year
  Occurrence of asthma exacerbation in 1 year after the study